CLINICAL TRIAL: NCT06945263
Title: Rectus Sheath Block and Coadministration of Intravenous Dexamethasone for Analgesia After Pediatric Laparoscopic Appendectomy - A Pilot Study
Brief Title: Comparing Pain Relief Between Two Methods of Freezing Injections in Children Having Their Appendix Removed
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: BC Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Prakash Krishnan, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H23-03547; F23-05308 (Other Grant/Funding Number: BC Children's Hospital Research Institute)
Record Dates: First submitted 2025-04-03; First posted 2025-04-25 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Laparoscopic Appendectomy
Keywords: Rectus Sheath Block; Dexamethasone; Laparoscopic Appendectomy; Analgesia; Anesthesia; Local Anesthetic
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectus Sheath Block with Intravenous Dexamethasone (Experimental): The rectus sheath block (RSB) is already current standard of care for laparoscopic appendectomy patients and is used by providers at the British Columbia Children's Hospital. The RSB group will receive up to a maximum of 1 mL/kg total of local anesthetic, which will ensure the total volume calculation for each arm will receive a bupivacaine dose at or below 2.5 mg/kg body weight. The anesthesia team will perform the bilateral RSBs using an in-plane ultrasound-guided technique with 0.25% bupivacaine with epinephrine 1:200 000 at 0.8 mL/kg (half of total volume per side) up to a maximum of 20 mL prior to the incision. The surgical team will then use the remaining 0.2 mL/kg to infiltrate the remaining port sites in RSB groups. Intravenous Dexamethasone will be administered concurrently.
  Interventions: Procedure: Rectus Sheath Block; Drug: Intravenous Dexamethasone; Drug: Local Anesthetic at the Incision Site
- Local Anesthetic (Active Comparator): Local anesthetic at the incision site is also current standard of care for appendectomy patients and is used by providers at the British Columbia Children's Hospital. This group will receive up to a maximum of 1 mL/kg total of LA which will ensure the total volume calculation for each arm would receive a bupivacaine dose at or below 2.5 mg/kg body weight. The local anesthetic infiltration arm will receive the same local anesthetic as the rectus sheath block arm (0.25% bupivacaine with epinephrine 1:200 000), injected by the surgeon. Surgeons can inject up to a total dose of 0.8 mL/kg (maximum 20 mL) at the umbilical port site. The remaining volume of local anesthetic (0.2 mL/kg) can be infiltrated at each of the incision sites at the discretion of the surgeon.
  Interventions: Drug: Local Anesthetic at the Umbilical Port Site; Drug: Local Anesthetic at the Incision Site

INTERVENTIONS:
Procedure: Rectus Sheath Block — Bilateral rectus sheath blocks using an in-plane ultrasound-guided technique with 0.25% bupivacaine with epinephrine 1:200 000 at 0.8 mL/kg (half of total volume per side) up to a maximum of 20 mL prior to the incision.
  Arms: Rectus Sheath Block with Intravenous Dexamethasone
Drug: Local Anesthetic at the Umbilical Port Site — 0.25% bupivacaine with epinephrine 1:200 000. Total dose of 0.8 mL/kg (maximum 20 mL) at the umbilical port site.
  Arms: Local Anesthetic
Drug: Intravenous Dexamethasone — Intravenous Dexamethasone delivered concurrent to the RSB. Total dose of 150 mcg/kg up to a maximum of 8 mg.
  Arms: Rectus Sheath Block with Intravenous Dexamethasone
Drug: Local Anesthetic at the Incision Site — The remaining volume of local anesthetic (0.2 mL/kg) can be infiltrated at each of the incision sites at the discretion of the surgeon up to a maximum of 10 mL.

SUMMARY:
Laparoscopic appendectomies are the most common emergency surgeries performed in children. Despite being considered minimally invasive surgeries, they can result in substantial postoperative pain and 2 of 3 patients require postoperative opioids. Increased postoperative pain can delay recovery, increase hospital admission time, lead to chronic pain, and cause patient distress. This study aims to reduce postoperative pain in this population by comparing the recovery outcomes associated with the administration of (1) an RSB with coadministration of IV dexamethasone as an LA adjunct (RSB+dex group) prior to the incision with (2) LA infiltration alone by the surgeon (LA group).

ELIGIBILITY:
Inclusion Criteria:

* Age 4-18 years old
* Diagnosed with acute appendicitis.
* Undergoing a laparoscopic appendectomy

Exclusion Criteria:

* Perforated/complicated appendicitis diagnosis
* Previous abdominal surgery
* Allergy to bupivacaine or dexamethasone
* Severe developmental delay preventing patients from using pain scales or adequately communicating pain
* Patients with Type 1 or 2 diabetes mellitus
* Patients with steroid dependence

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-04-27 (Estimated); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Total opioid administration | From the start of surgery until up to 16 hours post-operatively.
  Continuous variable measured by collecting and totaling all opioid (excluding remifentanil) administrations from intraoperative, anesthetic care unit (ACU), and ward records and converting to morphine milligram per kilogram equivalents.

SECONDARY OUTCOMES:
Mean postoperative pain score at 12 hours | 12 hours postoperatively
  Discrete variable measured via age-appropriate visual analog scale (Faces Pain Scale-Revised) for participants who are younger than 12 years old. The Faces Pain Scale is on a scale of 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Pain scores at 0 hours, 4 hours, 8 hours, and 16 hours postoperatively | 0 hours, 4 hours, 8 hours, and 16 hours postoperatively.
  Discrete variable measured via age-appropriate visual analog scale (FACES Pain Scale-Revised) for participants who are younger than 12 years old. The Faces Pain Scale is on a scale of 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time spent performing rectus sheath block | Intraoperatively.
  Time performing the rectus sheath block in minutes as recorded by the anesthesiologist.
Duration of anesthesia care unit (ACU) stay | Perioperatively.
  Time between ACU admission and discharge.
Duration of post-procedural hospitalization | Baseline (upon entering the operating room) to discharge from hospital, an average of 16 hours.
  Duration from entering the operating room to hospital discharge in minutes.
Parental perspective on patient postoperative pain | 24 to 72 hours postoperatively
  Parental assessment of patient postoperative pain using a numeric rating scale. The scale is from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Non-prescription postoperative drugs | 24 to 72 hours postoperatively
  Which non-prescription drugs are administered post-operatively from the parent to the patient.
Parental satisfaction with recovery | 24 to 72 hours postoperatively.
  Discrete 5-point scale (very unsatisfied, unsatisfied, neutral, satisfied, very satisfied) measuring parental satisfaction with patient recovery. Very unsatisfied is the worse outcome, very satisfied is the best outcome.
Mean Postoperative Pain Score at 12 Hours | 12 hours postoperatively
  Discrete variable measured via age-appropriate scale (Numeric Rating Scale) for participants who are 12 years old or older. The numeric rating scale is from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Pain scores at 0 hours, 4 hours, 8 hours, and 16 hours postoperatively | 0 hours, 4 hours, 8 hours, and 16 hours postoperatively.
  Discrete variable measured via age-appropriate scale (Numeric Rating Scale) for participants who are 12 years old or older. The numeric rating scale is from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Krishnan, MD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearson AME, Roberts S, Turbitt LR. New blocks on the kids: core basic nerve blocks in paediatric anaesthesia. Anaesthesia. 2023 Jan;78(1):3-8. doi: 10.1111/anae.15876. Epub 2022 Oct 11. No abstract available. PMID 36220155
- [Background] Shafy SZ, Miller R, Uffman JC, Tobias JD, Fetzer M, Nordin AB, Kenney B, Walia H, Veneziano G. An Enhanced Recovery Protocol that Facilitates Same-day Discharge for Simple Laparoscopic Appendectomies. Pediatr Qual Saf. 2019 Dec 5;4(6):e243. doi: 10.1097/pq9.0000000000000243. eCollection 2019 Nov-Dec. PMID 32010869
- [Background] Gee K, Ngo S, Burkhalter L, Beres AL. Safety and feasibility of same-day discharge for uncomplicated appendicitis: A prospective cohort study. J Pediatr Surg. 2018 May;53(5):988-990. doi: 10.1016/j.jpedsurg.2018.02.031. Epub 2018 Feb 9. PMID 29510871
- [Background] Cairo SB, Raval MV, Browne M, Meyers H, Rothstein DH. Association of Same-Day Discharge With Hospital Readmission After Appendectomy in Pediatric Patients. JAMA Surg. 2017 Dec 1;152(12):1106-1112. doi: 10.1001/jamasurg.2017.2221. PMID 28678998
- [Background] Alkhoury F, Burnweit C, Malvezzi L, Knight C, Diana J, Pasaron R, Mora J, Nazarey P, Aserlind A, Stylianos S. A prospective study of safety and satisfaction with same-day discharge after laparoscopic appendectomy for acute appendicitis. J Pediatr Surg. 2012 Feb;47(2):313-6. doi: 10.1016/j.jpedsurg.2011.11.024. PMID 22325382
- [Background] Cheng O, Cheng L, Burjonrappa S. Facilitating factors in same-day discharge after pediatric laparoscopic appendectomy. J Surg Res. 2018 Sep;229:145-149. doi: 10.1016/j.jss.2018.03.072. Epub 2018 Apr 25. PMID 29936981
- [Background] Pehora C, Pearson AM, Kaushal A, Crawford MW, Johnston B. Dexamethasone as an adjuvant to peripheral nerve block. Cochrane Database Syst Rev. 2017 Nov 9;11(11):CD011770. doi: 10.1002/14651858.CD011770.pub2. PMID 29121400
- [Background] Edinoff AN, Houk GM, Patil S, Bangalore Siddaiah H, Kaye AJ, Iyengar PS, Cornett EM, Imani F, Mahmoudi K, Kaye AM, Urman RD, Kaye AD. Adjuvant Drugs for Peripheral Nerve Blocks: The Role of Alpha-2 Agonists, Dexamethasone, Midazolam, and Non-steroidal Anti-inflammatory Drugs. Anesth Pain Med. 2021 Jul 4;11(3):e117197. doi: 10.5812/aapm.117197. eCollection 2021 Jun. PMID 34540647
- [Background] Desai N, Albrecht E. Local anaesthetic adjuncts for peripheral nerve blockade. Curr Opin Anaesthesiol. 2023 Oct 1;36(5):533-540. doi: 10.1097/ACO.0000000000001272. Epub 2023 Jun 14. PMID 37314172
- [Background] Maloney C, Kallis M, El-Shafy IA, Lipskar AM, Hagen J, Kars M. Ultrasound-guided bilateral rectus sheath block vs. conventional local analgesia in single port laparoscopic appendectomy for children with nonperforated appendicitis. J Pediatr Surg. 2018 Mar;53(3):431-436. doi: 10.1016/j.jpedsurg.2017.05.027. Epub 2017 Jun 2. PMID 28610706
- [Background] Hamill JK, Liley A, Hill AG. Rectus sheath block for laparoscopic appendicectomy: a randomized clinical trial. ANZ J Surg. 2015 Dec;85(12):951-6. doi: 10.1111/ans.12950. Epub 2015 Jan 12. PMID 25581711
- [Background] Hamill JK, Rahiri JL, Liley A, Hill AG. Rectus sheath and transversus abdominis plane blocks in children: a systematic review and meta-analysis of randomized trials. Paediatr Anaesth. 2016 Apr;26(4):363-71. doi: 10.1111/pan.12855. Epub 2016 Feb 4. PMID 26846889
- [Background] Russell P, von Ungern-Sternberg BS, Schug SA. Perioperative analgesia in pediatric surgery. Curr Opin Anaesthesiol. 2013 Aug;26(4):420-7. doi: 10.1097/ACO.0b013e3283625cc8. PMID 23756911
- [Background] Bosenberg A. Benefits of regional anesthesia in children. Paediatr Anaesth. 2012 Jan;22(1):10-8. doi: 10.1111/j.1460-9592.2011.03691.x. Epub 2011 Sep 7. No abstract available. PMID 21895855
- [Background] Yu TC, Hamill JK, Liley A, Hill AG. Warm, humidified carbon dioxide gas insufflation for laparoscopic appendicectomy in children: a double-blinded randomized controlled trial. Ann Surg. 2013 Jan;257(1):44-53. doi: 10.1097/SLA.0b013e31825f0721. PMID 22824858
- [Background] Shim H, Gan TJ. Side effect profiles of different opioids in the perioperative setting: are they different and can we reduce them? Br J Anaesth. 2019 Sep;123(3):266-268. doi: 10.1016/j.bja.2019.06.009. Epub 2019 Jul 17. No abstract available. PMID 31326087
- [Background] Tomecka MJ, Bortsov AV, Miller NR, Solano N, Narron J, McNaull PP, Ricketts KJ, Lupa CM, McLean SA. Substantial postoperative pain is common among children undergoing laparoscopic appendectomy. Paediatr Anaesth. 2012 Feb;22(2):130-5. doi: 10.1111/j.1460-9592.2011.03711.x. Epub 2011 Sep 29. PMID 21958060

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT06945263/Prot_SAP_000.pdf